CLINICAL TRIAL: NCT02453399
Title: Relief of Migraine Pain Through Transcutaneous Electro Stimulation
Brief Title: Relief of Migraine Pain Through Electro Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Theranica (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: RMB001115
Record Dates: First submitted 2015-05-13; First posted 2015-05-25 (Estimated); Last update posted 2017-12-08 (Actual); Status verified 2016-05

CONDITIONS: Migraine Headache
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Randomized treatment/placebo delivery of transcutaneous electro stimulation via a dedicated device Avital. — Transcutaneous electro stimulation

SUMMARY:
This study will evaluate transcutaneous electro stimulation device developed by Siano for adequacy, safety and efficacy for the treatment and/or prevention of migraine pain for migraine sufferers.

DETAILED DESCRIPTION:
This study will gather information regarding performance of Avital transcutaneous electro stimulation device developed by Siano. Electrostimulation in the form of weak electrical pulses arranged in specific patterns (programs), is delivered through adhesive electrodes attached to patient's skin. A set of stimulation programs, out of which one is placebo, is stored in device memory.The device is controlled wirelessly using a dedicated smartphone application. Participants will be instructed to attach and activate the device at the onset of a migraine attack and manually adjust stimulation intensity to a level where it is perceivable but not painful. Upon each activation, a program will be automatically picked for execution in random order. Randomization is performed within and between subjects. Subjects will not be aware of the executed program. Subjects are requested to refrain from use of migraine relief drugs prior to treatment and during the first two hours of the treated attack. Throughout the course of electrostimulation, participants will be requested to rate their migraine pain level via te same smartphone application, using Visual Analog Scale (VAS).

Overall experimental duration for each participant will be determined by the goal of using the Avital device for 10-20 migraine attacks.

Data containing activation times, executed programs, stimulation intensity and user feedback will be transmitted via the smartphone to a central database for analysis. All data are completely de-identified and linked to a unique code assigned to each device. The link between participant's ID and this code will be securely maintained by the research coordinator. Database will be overseen by Siano staff responsible for monitoring the clinical study. The electronic database will be used to generate outcome measures.

In the course of this study the investigators will obtain controlled data on the safety and efficacy of transcutaneous electro stimulation for migraine treatment using Siano developed transcutaneous electro stimulation device.

ELIGIBILITY:
Inclusion Criteria:

* Matches International Headache Society criteria for migraine with and without aura
* Reports 2-8 migraine attacks per month

Exclusion Criteria:

* Has other significant pain problem (e.g.cancer pain, fibromyalgia or other head or facial disorder) that in the opinion of the investigator may confound the study assessments
* Has severe cardiac or cerebrovascular disease
* Has uncontrolled high blood pressure (systolic >160 diastolic > 100 after 3 repeated measurements within 24 hours)
* Is currently implanted with an electrical and/or neurostimulator device (e.g. cardiac pacemaker or defibrillator, vagal neurostimulator, deep brain stimulator, spinal stimulator, bone growth stimulator cochlear implant, Sphenopalatine ganglion stimulator or Occipital nerve stimulator)
* Known epilepsy
* Use of Cannabis including medical use.
* Has chronic migraine (more than 15 headache days per month).
* Has undergone nerve block (occipital or other) in the head or neck within the last 2 months.
* Has received Botox injections within the last 6 months.
* Is pregnant or thinking of becoming pregnant during the study period, or of childbearing years and is unwilling to use an accepted form of birth control.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2015-07; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Migraine relief at 2 hours post treatment as determined by difference of reported pain levels at the beginning and 2 hours after the end of electro stimulation session. Pain levels are assessed by means of Numerical Pain Scale. | 2.5 hours
Relative migraine pain relief at 2 hours post treatment | 2.5 hours
  Relative migraine pain relief at 2 hours post treatment as determined by difference of reported pain levels at the beginning and 2 hours after the end of electro stimulation session normalized by pain level on start of the session. Pain levels are assessed by means of Numerical Pain Scale.
Percent responders resulted in significant pain relief at 2 hours post treatment | 2.5 hours
  Percent of responders with improvement of 50% or better in pain level according to NPS

SECONDARY OUTCOMES:
Migraine attack duration as determined by time between reported onset of migraine attack and time when, for this attack, reported pain level drops by at least three levels. Pain levels are assessed by means of Visual Analog Scale . | 2.5 hours
Use of pain relief medications as assessed by participants' reports at follow-up. | 6 months
  Use of pain relief medications, including dosage
Number of migraine attacks per month as determined by the number of activations. | 6 months
Overall wellbeing as assessed by means of post-study questionnaire | 6 months
Treatment related adverse effects, as assessed by means of post-study questionnaire, or participants' reports during the study. | 6 months
Migraine Relief at end of treatment as determined by difference of reported pain levels at the beginning of the electro stimulation and in the end of the electro stimulation session. Pain levels are assessed by means of NPS . | 0.5 hours

CONTACTS AND LOCATIONS:
Overall Officials: David Yarnitsky, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Medical Center, Haifa, Israel

REFERENCES:
- [Derived] Yarnitsky D, Volokh L, Ironi A, Weller B, Shor M, Shifrin A, Granovsky Y. Nonpainful remote electrical stimulation alleviates episodic migraine pain. Neurology. 2017 Mar 28;88(13):1250-1255. doi: 10.1212/WNL.0000000000003760. Epub 2017 Mar 1. PMID 28251920